CLINICAL TRIAL: NCT07254130
Title: COMPARISON OF MEAN DURATION OF POST OPERATIVE ANALGESIA FOLLOWING ADDITION OF DEXMEDETOMIDINE TO ROPIVACAINE VERSUS PLAIN ROPIVACAINE ON ULTRASOUND GUIDED RECTUS SHEATH BLOCK IN PATIENTS UNDERGOING MIDLINE LAPAROTOMIES
Brief Title: COMPARISON OF MEAN DURATION OF POST OPERATIVE ANALGESIA FOLLOWING ADDITION OF DEXMEDETOMIDINE TO ROPIVACAINE VERSUS PLAIN ROPIVACAINE ON ULTRASOUND GUIDED RECTUS SHEATH BLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Anam Mahmood, Principal investigator, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVH-2025-CT-012
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Midline Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine only group (Active Comparator)
  Interventions: Procedure: Rectus Sheath Block
- Dexmedetomedine combined with ropivacaine group (Active Comparator)
  Interventions: Procedure: Rectus Sheath Block

INTERVENTIONS:
Procedure: Rectus Sheath Block — In Dexmedetomedine combined with ropivacaine group, under ultrasound guidance, the needle will be advanced posterior to the rectus muscle, and 20 ml of 0.25% ropivacaine mixed with 1ug/kg body weight will be injected to hydrodissect the rectus muscle from the posterior sheath.
  In ropivacine only group, under ultrasound guidance, the needle will be advanced posterior to the rectus muscle, and 20 ml of 0.25% ropivacaine will be injected to hydrodissect the rectus muscle from the posterior sheath.

SUMMARY:
To compare the mean duration of postoperative analgesia following addition of dexmedetomidine to ropivacaine versus plain ropivacaine in ultrasound guided rectus sheath block in patients undergoing midline laparotomies

ELIGIBILITY:
Inclusion Criteria:

Patients with age 30 - 60 years.

* Patients that will be scheduled for laparotomy under general anesthesia.
* ASA (American Society of Anesthesiologist) s

Exclusion Criteria:

* Patient who will refuse for participation in study.
* Infection at site of Rectus Sheath block.
* History of any addiction.
* Sensitivity to the local anesthetics.
* Patient with pre-existing coagulation abnormalities INR more than 1.5.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Mean duration of analgesia | Baseline , 30 minutes , 2 hours, 4 hours , 6 hours , 8 hours , 12 hours , 24 hours
  Assessed using the visual analogue score(VAS) ranging from 0-10 (0=no pain , 10= most severe unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Bahawalpur, Punjab Province, Pakistan